CLINICAL TRIAL: NCT06423534
Title: Empowering New Mothers: Exploring the Effect of Breastfeeding Health Educational Program on Practices and Feeding Self-Efficacy of Primigravida in Saudi Arabia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-2024-126
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Primigravida Women

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study GROUP (Experimental): Each primigravida in the study group during the last three trimesters will receive three sessions of knowledge, breast care, and breastfeeding technique after filling out a questionnaire (pretest). During 1 month from delivery, we will conduct a post-test with them (after 2 weeks and after 4 weeks) to explore the effect of breastfeeding health educational programs on practices and breastfeeding self-efficacy
  Interventions: Behavioral: Breastfeeding Health Educational Program
- Control group (Active Comparator): The control group was selected first and received a brochure leaflet delivered by the researcher. They didn't receive the health educational program
  Interventions: Behavioral: Breastfeeding Health Educational Program

INTERVENTIONS:
Behavioral: Breastfeeding Health Educational Program — Breastfeeding is a mother's priceless gift to her infant and nature's own method of nurturing a baby. Therefore, this study will be conducted to evaluate the primigravida mother's breastfeeding's knowledge, attitude and corrective technique through the implementation of an educational program and to ascertain the efficacy of such a program.

SUMMARY:
Being pregnant causes a mother and her child to form a maternal tie, and the birth of the child fills the mother with an immense amount of love and happiness. Breastfeeding is how a mother and infant make their initial touch. Breastfeeding is a mother's priceless gift to her infant and nature's own method of nurturing a baby.

DETAILED DESCRIPTION:
This study will be done to evaluate the primigravida mother's breastfeeding's knowledge, attitude and corrective technique through the implementation of an educational program and to ascertain the efficacy of such a program.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida mothers who regularly visit maternity hospitals at Hail and Bisha City.
* Primigravida mothers during last three trimester and 1 month after delivery
* No problems during pregnant and have a healthy baby
* Primigravida mothers who are not contraindicated to breastfeeding

Exclusion Criteria:

* Multigravida mothers and pregnant women during first and second trimester

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
A preformatted structured questionnaire | 3 months
  It was developed by Tella et al. (2016) and comprised 12 questions that were assessed in various areas under various breastfeeding techniques practice.
Self-Efficacy Scale - Short-Form (BSES-SF) | 3 months
  It was adopted (Dennis, 2003) that assess maternal self-efficacy for breastfeeding throughout all stages of the study. The BSES-SF is a Likert scale with 14 items organized into two domains, namely: technical and intrapersonal thoughts.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Hail university, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No